CLINICAL TRIAL: NCT00003888
Title: A Randomized Phase III Multicenter Trial of Neoadjuvant Docetaxel (Taxotere) Plus Cisplatin Plus 5-Fluorouracil Versus Neoadjuvant Cisplatin Plus 5-Fluorouracil in Patients With Locally Advanced Inoperable Squamous Cell Carcinoma of the Head and Neck
Brief Title: Combination Chemotherapy Plus Radiation Therapy in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-24971; RP-56976-V-323
Record Dates: First submitted 1999-11-01; First posted 2004-01-29 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2015-07

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Docetaxel; Fluorouracil; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: fluorouracil
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug and combining chemotherapy with radiation therapy may kill more tumor cells. It is not yet known which regimen of combination chemotherapy is more effective for advanced head and neck cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of two regimens of combination chemotherapy plus radiation therapy in treating patients who have advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the progression free survival of patients with locally advanced, inoperable squamous cell carcinoma of the head and neck treated with cisplatin plus fluorouracil with or without docetaxel as a neoadjuvant to radiotherapy. II. Compare the response rate, response duration, toxicity, local symptoms, and time to disease progression of these treatment regimens in this patient population. III. Evaluate the quality of life in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to primary tumor site (oral cavity vs oropharynx vs hypopharynx vs larynx) and institution. Patients are randomized to one of two treatment arms. Arm I: Patients receive docetaxel IV over 1 hour, immediately followed by cisplatin IV over 1 hour on day 1 and fluorouracil (5-FU) IV as a continuous infusion on days 1-5. Arm II: Patients receive cisplatin IV over 1 hour on day 1 followed by 5-FU IV as a continuous infusion on days 1-5. Treatment continues every 3 weeks for 4 courses in the absence of disease progression or unacceptable toxicity. Patients receive radiotherapy following chemotherapy within 3-6 weeks of last course. Radiotherapy is administered 5 days a week for up to 7 weeks. Quality of life is assessed before treatment, at courses 2 and 4, and at 6 and 9 months. Patients are followed every 3 months for the first 2 years and then every 6 months until death.

PROJECTED ACCRUAL: A total of 348 patients will be accrued for this study within 24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven locally advanced squamous cell carcinoma of the head and neck Stage III or IV without distant metastases Unresectable Primary tumor sites: Oral cavity Oropharynx Hypopharynx Larynx Must have at least one measurable lesion

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than upper limit of normal (ULN) SGOT and SGPT no greater than 2.5 times ULN Alkaline phosphatase no greater than 5 times ULN No SGOT and SGPT greater than 1.5 times ULN AND alkaline phosphatase greater than 2.5 times ULN Renal: Creatinine no greater than 1.4 mg/dL OR Creatinine clearance at least 60 mL/min Cardiovascular: At least 6 months since prior myocardial infarction No unstable, treated cardiac disease Pulmonary: At least one year since prior hospitalization for chronic obstructive pulmonary disease Neurologic: No neurologic or psychiatric disorders (e.g., dementia or seizures) No concurrent peripheral neuropathy greater than grade 1 Other: No active uncontrolled infection No active peptic ulcer No alteration in hearing At least 5 years since any other neoplastic disease except curatively treated basal or squamous cell skin cancer, carcinoma in situ of the cervix, or other cancer curatively treated by surgery Not pregnant or nursing Fertile patients must use effective contraception No other psychological, familial, sociological, or geographical condition that would prevent compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: No primary prophylactic colony stimulating factors during the first course of therapy Chemotherapy: No prior or concurrent chemotherapy Endocrine therapy: At least 3 weeks since prior corticosteroid No chronic corticosteroid therapy (greater than 3 months) Radiotherapy: No prior radiotherapy Surgery: No prior surgery for this cancer Other: At least 30 days since prior treatment in a clinical trial No concurrent use of drugs that interact with fluorouracil (e.g., cimetidine, allopurinol, folic acid or leucovorin calcium) No other concurrent investigational drugs or anticancer treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 1999-04; Primary Completion 2002-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan B. Vermorken, MD, PhD, Study Chair — University Hospital, Antwerp
Locations (44):
- Austria (3):
  - Landeskrankenhaus/Universitatskliniken Graz, Graz
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (5):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Clinique Universitaire De Mont-Godinne, Mont-Godinne Yvoir
- Institute of Oncology and Radiology of Serbia, Belgrade, Federal Republic of Yugoslavia
- France (7):
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Oscar Lambret, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - CHR Hotel Dieu, Nantes
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
- Germany (3):
  - Martin Luther Universitaet, Halle
  - Caritasklinik St. Theresia, Saarbrücken
  - Mutterhaus der Borromaerinnen, Trier
- Ahepa University Hospital, Thessaloniki, Greece
- Hungary (3):
  - National Institute of Oncology, Budapest
  - Szent Margit Hospital, Budapest
  - Borsod-Abauj-Zemplen County Hospital, Miskolc
- Italy (4):
  - Centro di Riferimento Oncologico - Aviano, Aviano
  - Ospedale Santa Croce, Cuneo
  - Istituti Fisioterapici Ospitalieri - Roma, Rome
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (4):
  - Academisch Medisch Centrum, Amsterdam
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - University Medical Center Nijmegen, Nijmegen
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- National Cancer Institute - Bratislava, Bratislava, Slovakia
- Spain (4):
  - Institut Catala d'Oncologia - Hospital Duran i Reynals, Barcelona
  - Hospital General de Jerez, Jerez de la Frontera
  - Universidad de Santiago - Hospital de Conxo, Santiago de Compostela
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (2):
  - Kantonspital Aarau, Aarau
  - Ospedale San Giovanni, Bellinzona
- Istanbul University-Institute of Oncology, Istanbul, Turkey (Türkiye)
- United Kingdom (4):
  - Charing Cross Hospital, London, England
  - Middlesex Hospital- Meyerstein Institute, London, England
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Beatson Oncology Centre, Glasgow, Scotland

REFERENCES:
- [Background] Jansen J, Vermorken JB, Boote D, et al.: Cost-effectiveness analysis of the EORTC 24971 (TAX 323) trial comparing docetaxel plus cisplatin and 5-fluorouracil versus standard treatment (cisplatin and 5-fluorouracil) as induction chemotherapy followed by radiation therapy in locally advanced unresectable squamous cell carcinoma of the head and neck (SCCHN). [Abstract] J Clin Oncol 25 (Suppl 18): A-6090, 321s, 2007.
- [Result] van Herpen CM, Mauer ME, Mesia R, Degardin M, Jelic S, Coens C, Betka J, Bernier J, Remenar E, Stewart JS, Preiss JH, van den Weyngaert D, Bottomley A, Vermorken JB; EORTC Head and Neck Group. Short-term health-related quality of life and symptom control with docetaxel, cisplatin, 5-fluorouracil and cisplatin (TPF), 5-fluorouracil (PF) for induction in unresectable locoregionally advanced head and neck cancer patients (EORTC 24971/TAX 323). Br J Cancer. 2010 Oct 12;103(8):1173-81. doi: 10.1038/sj.bjc.6605860. Epub 2010 Sep 14. PMID 20842129
- [Result] Vermorken JB, Remenar E, van Herpen C, Gorlia T, Mesia R, Degardin M, Stewart JS, Jelic S, Betka J, Preiss JH, van den Weyngaert D, Awada A, Cupissol D, Kienzer HR, Rey A, Desaunois I, Bernier J, Lefebvre JL; EORTC 24971/TAX 323 Study Group. Cisplatin, fluorouracil, and docetaxel in unresectable head and neck cancer. N Engl J Med. 2007 Oct 25;357(17):1695-704. doi: 10.1056/NEJMoa071028. PMID 17960012
- [Result] Bernier J, Coens C, Remenar E, et al.: Impact on quality of life (QoL) of the addition of docetaxel (T) to neoadjuvant cisplatin plus 5-fluorouracil treatment in patients with locally advanced unresectable squamous cell carcinoma of the head and neck (SCCHN): EORTC study 24971. [Abstract] J Clin Oncol 24 (Suppl 18): A-5522, 285s, 2006.
- [Result] Remenar E, Van Herpen C, Lluch JG, et al.: A randomized phase III multicenter trial of neoadjuvant docetaxel plus cisplatin and 5-fluorouracil (TPF) versus neoadjuvant PF in patients with locally advanced unresectable squamous cell carcinoma of the head and neck (SCCHN). Final analysis of EORTC 24971. [Abstract] J Clin Oncol 24 (Suppl 18): A-5516, 2006.
- [Result] Vermorken JB, Remenar E, Van Herpen C, et al.: Standard cisplatin/infusional 5-fluorouracil (PF) vs docetaxel (T) plus PF (TPF) as neoadjuvant chemotherapy for nonresectable locally advanced squamous cell carcinoma of the head and neck (LA-SCCHN): a phase III trial of the EORTC Head and Neck Cancer Group (EORTC #24971). [Abstract] J Clin Oncol 22 (Suppl 14): A-5508, 490s, 2004.